CLINICAL TRIAL: NCT04641585
Title: Brugada Syndrome and Artificial Intelligence Applications to Diagnosis
Acronym: BrAID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto di Fisiologia Clinica CNR (Other)
Collaborators: Fondazione Toscana Gabriele Monasterio (Other); Azienda USL Toscana Sud Est (Other Government); Azienda USL Toscana Nord Ovest (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BrAID
Record Dates: First submitted 2020-10-22; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Brugada Syndrome 1
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients affected by Brugada Syndrome 1 (Experimental): Patients with spontaneous or drug-induced Brugada Syndrome 1
  Interventions: Diagnostic Test: Patients affected by Brugada Syndrome 1
- Controls (Active Comparator): Patients with no condition associated with spontaneous or drug-induced Brugada Syndrome 1
  Interventions: Diagnostic Test: Patients affected by Brugada Syndrome 1

INTERVENTIONS:
Diagnostic Test: Patients affected by Brugada Syndrome 1 — ECG analysis by Machine Learning algorithms and blood collection for the transcriptomic study of markers possibly associated with the disease

SUMMARY:
Aim of the project is the development of an integrated platform, based on machine learning and omic techniques, able to support physicians in as much as possible accurate diagnosis of Type 1 Brugada Syndrome (BrS).

DETAILED DESCRIPTION:
The aim of BrAID project is to integrate classic clinical guidelines for Brugada Syndrome 1 diagnosis evaluation with innovative Information and Communication Technologies and omic approaches, generating new diagnostic strategies in cardiovascular precision medicine of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Brugada patients: patients with Brugada Syndrome 1 spontaneous or induced by the ajmaline test; patients with non-diagnostic electrocardiographic pattern for Brugada Syndrome 1 or negative in the presence of high clinical suspicion (family history for Brugada Syndrome, patients who survived cardiac arrest without organic heart disease)
* Control patients: patients with frequent premature ventricular complex and normal left and right ventricular function; patients with suspected Brugada Syndrome 1 not confirmed by ajmaline test

Exclusion Criteria:

* organic heart disease or diseases interfering with protocol completion
* lack of signed informed consent
* pregnancy
* acute coronary artery disease, heart failure in the previous 3 months
* severe renal or liver failure

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Machine Learning recognition of Brugada Syndrome 1 | Week 20
  Identification of Brugada type 1 Syndrome coved ST component in a cohort of 44 patients (prospective study) and validated in a cohort of 100 patients (validation study) according to the diagnostic patterns related to Brugada Syndrome 1 on 12-leads ECG as already published on current international guidelines
Machine Learning recognition of Brugada Syndrome 1 | Week 20
  Identification of Brugada type 1 Syndrome QRS fragmentation component in a cohort of 44 patients (prospective study) and validated in a cohort of 100 patients (validation study) according to the diagnostic patterns related to Brugada Syndrome 1 on 12-leads ECG as already published on current international guidelines
Machine Learning recognition of Brugada Syndrome 1 | Week 20
  Identification and characterization of Brugada type 1 Syndrome T segment depression component in a cohort of 44 patients (prospective study) and validated in a cohort of 100 patients (validation study) according to the diagnostic patterns related to Brugada Syndrome 1 on 12-leads ECG as already published on current international guidelines
Machine Learning recognition of Brugada Syndrome 1 | Week 20
  Identification of Brugada type 1 Syndrome broad P wave with PQ prolongation component in a cohort of 44 patients (prospective study) and validated in a cohort of 100 patients (validation study) according to the diagnostic patterns related to Brugada Syndrome 1 on 12-leads ECG as already published on current international guidelines

SECONDARY OUTCOMES:
Biomarkers associated with Brugada Syndrome 1 | week 48
  Identification of biomarkers associated with Brugada Syndrome 1 by the means of blood transcriptomic profile and exosomes analysis of patients. Transcriptomic and exosome could provide new insight into the pathophysiology of signalling in this pathology, as well as for application in Brugada Syndrome 1 diagnosis and therapeutics.
  Transcriptomic will provide a global picture of phenotypical changes associated with the disease, highlighting the potential genes involved in the development of Brugada Syndrome 1 The analysis of exosome coding and noncoding RNAs, participating in a variety of basic cellular functions, could also evidence potentially important pathophysiologic effects both in cardiac cells as well as on the release of electrical stimuli.
  The study will be performed in a cohort of 44 patients (prospective study) and results will be validated in a cohort of 100 patients (validation study)
Stratification risk | week 64
  Development of stratification risk system for Brugada type 1 Syndrome by the integration of ECG Machine Learning algorithms and biomarkers. In particular, the module will combine the peculiar ECG patterns associated with BrS (coved ST, QRS fragmentation, T segment depression, broad P wave with PQ prolongation)(outcome 1-4) and omic (genes) and exosome markers (coding and noncoding RNAs)(outcome 5) with the aim to improve patient risk stratification.
  Specifically, gene expression modulation (expressed as % respect to control population) of Na+ (e.g., Nav1.5, Nav1.3, Nav2.1), Ca2+ (e.g. Cav3.1, HCN3) and K+ channels (e.g.,TWIK1, Kv4.3) will be evaluated.
  The study will be performed in a cohort of 44 patients (prospective study) and results will be validated in a cohort of 100 patients (validation study).

CONTACTS AND LOCATIONS:
Overall Officials: Federico Vozzi, Ph.D., Principal Investigator — Istituto di Fisiologia Clinica
Locations (6):
- Italy (6):
  - Azienda USL Toscana Sud Est - U.O.C Cardiologia, Arezzo, Tuscany
  - Azienda Ospedaliera Universitaria Careggi - SOD Aritmologia, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana - Cardiologia 2, Pisa, Tuscany
  - Fondazione Toscana Gabriele Monasterio, Pisa, Tuscany
  - Istituto di Fisiologia Clinica IFC-CNR, Pisa, Tuscany
  - Azienda Usl Toscana Nord Ovest - U.O.C. Cardiologia, Viareggio, Tuscany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brugada P, Brugada J. Right bundle branch block, persistent ST segment elevation and sudden cardiac death: a distinct clinical and electrocardiographic syndrome. A multicenter report. J Am Coll Cardiol. 1992 Nov 15;20(6):1391-6. doi: 10.1016/0735-1097(92)90253-j. PMID 1309182
- [Background] Quan XQ, Li S, Liu R, Zheng K, Wu XF, Tang Q. A meta-analytic review of prevalence for Brugada ECG patterns and the risk for death. Medicine (Baltimore). 2016 Dec;95(50):e5643. doi: 10.1097/MD.0000000000005643. PMID 27977610
- [Background] Vutthikraivit W, Rattanawong P, Putthapiban P, Sukhumthammarat W, Vathesatogkit P, Ngarmukos T, Thakkinstian A. Worldwide Prevalence of Brugada Syndrome: A Systematic Review and Meta-Analysis. Acta Cardiol Sin. 2018 May;34(3):267-277. doi: 10.6515/ACS.201805_34(3).20180302B. PMID 29844648
- [Background] Antzelevitch C, Brugada P, Borggrefe M, Brugada J, Brugada R, Corrado D, Gussak I, LeMarec H, Nademanee K, Perez Riera AR, Shimizu W, Schulze-Bahr E, Tan H, Wilde A. Brugada syndrome: report of the second consensus conference. Heart Rhythm. 2005 Apr;2(4):429-40. doi: 10.1016/j.hrthm.2005.01.005. PMID 15898165
- [Background] Wilde AA, Antzelevitch C, Borggrefe M, Brugada J, Brugada R, Brugada P, Corrado D, Hauer RN, Kass RS, Nademanee K, Priori SG, Towbin JA; Study Group on the Molecular Basis of Arrhythmias of the European Society of Cardiology. Proposed diagnostic criteria for the Brugada syndrome. Eur Heart J. 2002 Nov;23(21):1648-54. doi: 10.1053/euhj.2002.3382. No abstract available. PMID 12448445
- [Background] Sarquella-Brugada G, Campuzano O, Arbelo E, Brugada J, Brugada R. Brugada syndrome: clinical and genetic findings. Genet Med. 2016 Jan;18(1):3-12. doi: 10.1038/gim.2015.35. Epub 2015 Apr 23. PMID 25905440
- [Derived] Morales MA, Piacenti M, Nesti M, Solarino G, Pieragnoli P, Zucchelli G, Del Ry S, Cabiati M, Vozzi F. The BrAID study protocol: integration of machine learning and transcriptomics for brugada syndrome recognition. BMC Cardiovasc Disord. 2021 Oct 13;21(1):494. doi: 10.1186/s12872-021-02280-3. PMID 34645390